CLINICAL TRIAL: NCT05740267
Title: Natural Orifice Specimen Extraction Surgery for Colorectal Cancer (NOSE for CRC)
Brief Title: Natural Orifice Specimen Extraction Surgery for Colorectal Cancer
Acronym: NOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102468A3
Record Dates: First submitted 2023-01-30; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization will be performed in the operating room at the Colorectal division, Linkou Chang Gung Memorial Hospital. Following the induction of minimally invasive surgery, an independent research assistant randomly assigned patients to undergo either NOSE surgery or conventional laparoscopic mini-laparotomy resection by sealed-envelope randomization.
Who Masked: Investigator
Masking Description: Randomization assignment is performed by the statisticians of the clinical trial center to generate random codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional laparoscopy group (No Intervention): The investigators can select either the intracorporeal or extracorporeal method to create bowel anastomoses. For the extracorporeal way, a mini-laparotomy wound is created and exteriorizes the bowel to do the anastomosis. The specimen is removed via the mini-laparotomy wound after the anastomosis is accomplished for the intracorporeal approach.
- NOSE group (Experimental): After bowel resection, all bowel anastomoses are created via side-to-side intracorporeal anastomosis, either isoperistaltic or antiperistaltic. The surgical steps of NOSE with the transrectal method are illustrated in Figure 1. First, the rectosigmoid colonic lumen is blocked with a bowel clamp. After rectal irrigation with povidone-iodine water, a transanal endoscopic microsurgery (TEM) scope or Alexis wound protector is inserted through the anus, reaching the upper rectum. Enterotomy is performed at the upper rectum, and a suction device is used to clean any fecal spillage. The TEM scope is pushed forward beyond the rectal opening, and the specimen is extracted with the TEM scope. The rectal opening is closed with a barbed suture, and an air leak test is performed to identify anastomotic leakage.
  Interventions: Procedure: Natural Orifice Specimen Extraction

INTERVENTIONS:
Procedure: Natural Orifice Specimen Extraction — After bowel resection, all bowel anastomoses are created via side-to-side intracorporeal anastomosis, either isoperistaltic or antiperistaltic. The surgical steps of NOSE with the transrectal method are illustrated in Figure 1. First, the rectosigmoid colonic lumen is blocked with a bowel clamp. After rectal irrigation with povidone-iodine water, a transanal endoscopic microsurgery (TEM) scope or Alexis wound protector is inserted through the anus, reaching the upper rectum. Enterotomy is performed at the upper rectum, and a suction device is used to clean any fecal spillage. The TEM scope is pushed forward beyond the rectal opening, and the specimen is extracted with the TEM scope. The rectal opening is closed with a barbed suture, and an air leak test is performed to identify anastomotic leakage.
  Arms: NOSE group

SUMMARY:
The goal of this type of study: a prospective, randomized controlled clinical trial is to assess the safety and feasibility of NOSE surgery to compare the NOSE and conventional laparoscopy groups in Colorectal cancer patients. The main questions it aims to answer are measuring the postoperative inflammatory response and monitoring the early morbidity and mortality rate after surgery. Participants will be assigned patients to undergo either NOSE surgery or conventional laparoscopic mini-laparotomy resection. If there is a comparison group: Researchers will compare the control group to see if postoperative inflammatory response.

DETAILED DESCRIPTION:
Endpoints (Outcome measure)：

Primary endpoint:

The primary outcome measure was the postoperative inflammatory response, which was evaluated by monitoring the C-reactive protein (CRP) level during hospitalization on the 3rd day following surgery. Early morbidity and mortality rate (postoperative 30 days): The early morbidity and mortality rate is defined as the event observed during the operation and within 30 days after surgery. Postoperative 30-day hospital readmission data will be also collected.

1. Secondary endpoints:

   A. Duration of Operation time: The length of the surgery will be recorded. B.Peritoneal Cytologyduring surgery: The investigators assess the tumor cells identified by peritoneal cytologic specimens. Given the relationship of positive cytology with metachronous peritoneal seeding, it is essential to evaluate datasets from patients who undergo the NOSE group.

   C. Peritoneal Contamination during surgery: Peritoneal fluid samples were collected under sterile circumstances at the end of the surgery and sent for aerobic and anaerobic cultures. The investigators evaluate the contamination rate of peritoneal fluid in the two groups.

   D.Postoperative Pain Score:

   Pain intensity is assessed using a Numeric Rating Scale (NRS) with scores from 0 to 10 (10 = the worst pain). The highest pain scores of patients on each day for three consecutive days postoperatively will be recorded for further evaluation.

   E.Postoperative Recovery course:

   Time to first flatus passage Time to the first liquid diet Time to the first soft diet The length of hospital stays F.Number of retrieved lymph nodes G.Recurrence incidence and pattern
2. Exploratory endpoints (if any):

Long-term outcome:

Overall survival Disease-free survival Cancer-specific survival Inclusion/Exclusion Criteria： Patient Enrollment Histological or cytological confirmation of colorectal adenocarcinoma. Inclusion criteria

1. Age ≥ 18
2. Performance status of 0 - 2 on the ECOG (Eastern Cooperative Oncology Group) scale
3. American Society of Anesthesiology (ASA) score is Ⅰ-Ⅲ
4. Tumor location: CRC with the lower margin of the tumor greater than 10 cm from the anal verge
5. Pre-operative T staging: T0-T4a at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
6. Preoperative M staging: M0 according to AJCC 8th
7. Tumor size: 4 cm or less
8. Written informed consent for participation Exclusion criteria

(1) Not suitable for minimally invasive surgery (2) Body mass index (BMI) >30 kg/m2 (3) Malnutrition: albumin level less than 3.5 (4) Previous pelvic surgery (5) Emergency surgery Study Procedures： Randomization Randomization will be performed in the operating room at the Colorectal division, Linkou Chang Gung Memorial Hospital. Following the induction of minimally invasive surgery, an independent research assistant randomly assigned patients to undergo either NOSE surgery or conventional laparoscopic mini-laparotomy resection by sealed-envelope randomization. To ensure every group is similar in terms of covariates, especially the operation method (including right hemicolectomy, left hemicolectomy, and anterior resection). Randomization assignment is performed by the statisticians of the clinical trial center to generate random codes.

Minimally invasive surgery Minimally invasive surgery will be performed in all operations, including multi-port laparoscopic surgery and robotic surgery. After the segment of bowel resection, the strategy for surgical specimen removal is according to the result of randomization.

# Conventional laparoscopy group: The investigators can select either the intracorporeal or extracorporeal method to create bowel anastomoses. For the extracorporeal way, a mini-laparotomy wound is created and exteriorizes the bowel to do the anastomosis. The specimen is removed via the mini-laparotomy wound after the anastomosis is accomplished for the intracorporeal approach.

# NOSE group: After bowel resection, all bowel anastomoses are created via side-to-side intracorporeal anastomosis, either isoperistaltic or antiperistaltic. The surgical steps of NOSE with the transrectal method are illustrated in Figure 1. First, the rectosigmoid colonic lumen is blocked with a bowel clamp. After rectal irrigation with povidone-iodine water, a transanal endoscopic microsurgery (TEM) scope or Alexis wound protector is inserted through the anus, reaching the upper rectum. Enterotomy is performed at the upper rectum, and a suction device is used to clean any fecal spillage. The TEM scope is pushed forward beyond the rectal opening, and the specimen is extracted with the TEM scope. The rectal opening is closed with a barbed suture, and an air leak test is performed to identify anastomotic leakage.

Intra-operative evaluation

Peritoneal lavage with 50 ml of normal saline on the Douglas pouch and the sub-phrenic area will be performed after the bowel anastomosis and before the abdominal wound closure. The estimated time would be 5 to 10 minutes. No additional risk will occur during the procedure. The investigators will do the peritoneal lavage fluid analysis in the following two phases:

* Peritoneal washing cytology (PWC) Peritoneal washing cytology (PWC) is a helpful indicator of peritoneal surface involvement and peritoneal dissemination of colorectal cancer. It may identify subclinical peritoneal spread and thus provide prognostic information. PWC is a useful prognostic tool in patients undergoing curative surgery for colorectal cancer since positive PWC was shown to be a potential risk factor for recurrence. The investigators will compare the positive rate of peritoneal cytology in the two groups.
* Peritoneal fluid bacterial culture:

Although minimally invasive surgery is performed with standard procedure, contamination is inconceivable to avoid. In the NOSE group, the rectum is opened and exposed to the peritoneal cavity, and bacterial contamination is inevitable. After finishing the anastomosis in each group, a microbiological sample is obtained from the peritoneal fluid specimens. The investigators will collect the data and analyze the correlation between NOSE and wound infection and intra-abdominal infection rates.

Post-operative assessment

The postoperative outcome will be analyzed as below:

1. Postoperative complications The complication within 30 days will be recorded and categorized according to the Clavien-Dindo classification.
2. Bowel function recovery The investigators will record and analyze the time to the first flatus passage, the first liquid diet, and the time to a soft diet.
3. The length of hospital stays The length of hospital stays is calculated from the date of operation to the discharge date.
4. Second operation and Readmission Reoperation and unplanned readmission will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Patient Enrollment Histological or cytological confirmation of colorectal adenocarcinoma. Inclusion criteria

1. Age ≥ 18
2. Performance status of 0 - 2 on the ECOG (Eastern Cooperative Oncology Group) scale
3. American Society of Anesthesiology (ASA) score is Ⅰ-Ⅲ
4. Tumor location: CRC with the lower margin of the tumor greater than 10 cm from the anal verge
5. Pre-operative T staging: T0-T4a at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition
6. Preoperative M staging: M0 according to AJCC 8th
7. Tumor size: 4 cm or less
8. Written informed consent for participation

Exclusion Criteria:

1. Not suitable for minimally invasive surgery
2. Body mass index (BMI) >30 kg/m2
3. Malnutrition: albumin level less than 3.5
4. Previous pelvic surgery
5. Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein (CRP) level | 3 minutes
  The primary outcome measure was the postoperative inflammatory response, which was evaluated by monitoring the C-reactive protein (CRP) level during hospitalization on the 3rd day following surgery. Complete blood cell count and differential count, C-reactive protein, procalcitonin, and interleukin-6 will be measured on day 3 postoperatively

SECONDARY OUTCOMES:
Duration of Operation time | 60~90 minutes
  The length of the surgery will be recorded.
Peritoneal Cytology during surgery | 3 minutes
  The investigators assess the tumor cells identified by peritoneal cytologic specimens. Given the relationship of positive cytology with metachronous peritoneal seeding, it is essential to evaluate datasets from participants who undergo the NOSE group. The investigators will compare the positive rate of peritoneal cytology in the two groups.
Peritoneal Contamination during surgery | 3 minutes
  Peritoneal fluid samples were collected under sterile circumstances at the end of the surgery and sent for aerobic and anaerobic cultures. The investigators evaluate the contamination rate of peritoneal fluid in the two groups. After finishing the anastomosis in each group, a microbiological sample is obtained from the peritoneal fluid specimens. The investigators will collect the data and analyze the correlation between NOSE and wound infection and intra-abdominal infection rates.
Postoperative Pain Score | 3 minutes
  Pain intensity is assessed using a Numeric Rating Scale (NRS) with scores from 0 to 10 (10 = the worst pain). The highest pain scores of patients on each day for three consecutive days postoperatively will be recorded for further evaluation.
Postoperative Recovery course: | 1 to 5 days
  Time to first flatus passage Time to first liquid diet Time to first soft diet The length of hospital stays

CONTACTS AND LOCATIONS:
Overall Officials: Jeng-Fu You, Study Director — Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu HM, Jen GH, Wang YW, Fann JC, Hsu CY, Jeng YC, Yen AM, Chiu SY, Chen SL, Hsu WF, Lee YC, Wu MS, Wu CY, Jou YY, Chen TH. Long-term effectiveness of faecal immunochemical test screening for proximal and distal colorectal cancers. Gut. 2021 Dec;70(12):2321-2329. doi: 10.1136/gutjnl-2020-322545. Epub 2021 Jan 25. PMID 33495268
- [Background] Clinical Outcomes of Surgical Therapy Study Group; Nelson H, Sargent DJ, Wieand HS, Fleshman J, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Ota D. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med. 2004 May 13;350(20):2050-9. doi: 10.1056/NEJMoa032651. PMID 15141043
- [Background] Green BL, Marshall HC, Collinson F, Quirke P, Guillou P, Jayne DG, Brown JM. Long-term follow-up of the Medical Research Council CLASICC trial of conventional versus laparoscopically assisted resection in colorectal cancer. Br J Surg. 2013 Jan;100(1):75-82. doi: 10.1002/bjs.8945. Epub 2012 Nov 6. PMID 23132548
- [Background] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061
- [Background] Kehlet H, Wilmore DW. Evidence-based surgical care and the evolution of fast-track surgery. Ann Surg. 2008 Aug;248(2):189-98. doi: 10.1097/SLA.0b013e31817f2c1a. PMID 18650627
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Scott MJ, Baldini G, Fearon KC, Feldheiser A, Feldman LS, Gan TJ, Ljungqvist O, Lobo DN, Rockall TA, Schricker T, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 1: pathophysiological considerations. Acta Anaesthesiol Scand. 2015 Nov;59(10):1212-31. doi: 10.1111/aas.12601. Epub 2015 Sep 8. PMID 26346577
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Saad S, Hosogi H. Natural orifice specimen extraction for avoiding laparotomy in laparoscopic left colon resections: a new approach using the McCartney tube and the tilt top anvil technique. J Laparoendosc Adv Surg Tech A. 2010 Oct;20(8):689-92. doi: 10.1089/lap.2010.0303. PMID 20874237
- [Background] Wolthuis AM, de Buck van Overstraeten A, Fieuws S, Boon K, D'Hoore A. Standardized laparoscopic NOSE-colectomy is feasible with low morbidity. Surg Endosc. 2015 May;29(5):1167-73. doi: 10.1007/s00464-014-3784-3. Epub 2014 Aug 23. PMID 25149636
- [Background] Park JS, Choi GS, Kim HJ, Park SY, Jun SH. Natural orifice specimen extraction versus conventional laparoscopically assisted right hemicolectomy. Br J Surg. 2011 May;98(5):710-5. doi: 10.1002/bjs.7419. Epub 2011 Feb 8. PMID 21305535
- [Background] Wolthuis AM, Fieuws S, Van Den Bosch A, de Buck van Overstraeten A, D'Hoore A. Randomized clinical trial of laparoscopic colectomy with or without natural-orifice specimen extraction. Br J Surg. 2015 May;102(6):630-7. doi: 10.1002/bjs.9757. Epub 2015 Mar 12. PMID 25764376
- [Background] Senft JD, Droscher T, Gath P, Muller PC, Billeter A, Muller-Stich BP, Linke GR. Inflammatory response and peritoneal contamination after transrectal natural orifice specimen extraction (NOSE) versus mini-laparotomy: a porcine in vivo study. Surg Endosc. 2018 Mar;32(3):1336-1343. doi: 10.1007/s00464-017-5811-7. Epub 2017 Aug 25. PMID 28842761
- [Background] Franklin ME Jr, Liang S, Russek K. Natural orifice specimen extraction in laparoscopic colorectal surgery: transanal and transvaginal approaches. Tech Coloproctol. 2013 Feb;17 Suppl 1:S63-7. doi: 10.1007/s10151-012-0938-y. Epub 2012 Dec 19. PMID 23250638
- [Background] Cheng CC, Hsu YR, Chern YJ, Tsai WS, Hung HY, Liao CK, Chiang JM, Hsieh PS, You JF. Minimally invasive right colectomy with transrectal natural orifice extraction: could this be the next step forward? Tech Coloproctol. 2020 Nov;24(11):1197-1205. doi: 10.1007/s10151-020-02282-x. Epub 2020 Jul 6. PMID 32632708
- [Background] Jong BK, Cheng CC, Hsu YJ, Chern YJ, Tsai WS, Hung HY, Liao CK, Yeh CY, Hsieh PS, You JF. Transrectal natural orifice specimen extraction in left hemicolectomy for tumours around the splenic flexure: Old wine in new bottles. Colorectal Dis. 2022 Jan;24(1):128-132. doi: 10.1111/codi.15930. Epub 2021 Oct 10. PMID 34601777
- [Background] Zhou ZQ, Wang K, Du T, Gao W, Zhu Z, Jiang Q, Ji F, Fu CG. Transrectal Natural Orifice Specimen Extraction (NOSE) With Oncological Safety: A Prospective and Randomized Trial. J Surg Res. 2020 Oct;254:16-22. doi: 10.1016/j.jss.2020.03.064. Epub 2020 May 8. PMID 32402832
- [Background] Muller PC, Dube A, Steinemann DC, Senft JD, Gehrig T, Benner L, Nickel F, Muller-Stich BP, Linke GR. Contamination After Disinfectant Rectal Washout in Left Colectomy as a Model for Transrectal NOTES: A Randomized Controlled Trial. J Surg Res. 2018 Dec;232:635-642. doi: 10.1016/j.jss.2018.07.066. Epub 2018 Aug 16. PMID 30463785
- [Background] Homma Y, Hamano T, Akazawa Y, Otsuki Y, Shimizu S, Kobayashi H, Kameoka S, Kobayashi Y. Positive peritoneal washing cytology is a potential risk factor for the recurrence of curatively resected colorectal cancer. Surg Today. 2014 Jun;44(6):1084-9. doi: 10.1007/s00595-013-0689-z. Epub 2013 Aug 14. PMID 23942820
- [Background] Salamanca IMG, Jaime MTE, Penco JMM, Martinez JS. Role of Peritoneal Cytology in Patients with Early Stage Colorectal Cancer. Pathol Oncol Res. 2020 Apr;26(2):1325-1329. doi: 10.1007/s12253-019-00706-0. Epub 2019 Aug 10. PMID 31401769
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Lo AL, Hsu YJ, Chern YJ, Cheng CC, Jong BK, Yu ZH, Chan LY, You JF; NOSE study group of Taiwan Colorectal Action Research Society. Mini-laparotomy versus transrectal natural orifice specimen extraction for minimally invasive colorectal cancer surgery: study protocol for a randomized controlled trial (MINITR-NOSE trial, TCAR2514 protocol). Trials. 2025 Aug 25;26(1):304. doi: 10.1186/s13063-025-09039-7. PMID 40855494